CLINICAL TRIAL: NCT00655798
Title: Effect of Nutritional Interventions on Inflammatory Status in Healthy Overweight Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Novonesis (Industry)
Responsible Party: Dr. G.C.M. Bakker, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P6957
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Overweight; Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Overweight; Diabetes Mellitus; Cardiovascular Diseases

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator)
  Interventions: Dietary Supplement: Plain Yogurt + mix of anti-oxidants capsules
- 3 (Active Comparator)
  Interventions: Dietary Supplement: Yogurt containing Lactobacillus helveticus
- 4 (Active Comparator)
  Interventions: Dietary Supplement: Yogurt containing Bifidobacterium animalis ssp.

INTERVENTIONS:
Dietary Supplement: Placebo — plain yogurt and capsules containing cellulose
  Arms: 1
Dietary Supplement: Plain Yogurt + mix of anti-oxidants capsules — plain yogurt and capsules containing mix of anti-oxidants
  Arms: 2
Dietary Supplement: Yogurt containing Lactobacillus helveticus — Yogurt containing the probiotic Lactobacillus helveticus
  Arms: 3
Dietary Supplement: Yogurt containing Bifidobacterium animalis ssp. — Yogurt containing the probiotic Bifidobacterium animalis ssp.
  Arms: 4

SUMMARY:
In the present study it is hypothesized that a reduction of the inflammatory status may prevent the occurrence of disorders and diseases related to overweight.

In this study the effects of nutritional compounds will be studied in overweight men with a low grade inflammatory status. We will investigate the effects of 3 different food treatments as compared to a placebo on markers of inflammation and on parameters of glucose and fat metabolism. The three different food treatments are a food mix and two yogurts each containing different probiotic strains. The food mix is composed of a mix of nutritional components, each reported to affect inflammation parameters and (or) anti-oxidant status but different in their -hypothesized-mode of action.

DETAILED DESCRIPTION:
From day -01 onwards until the end of the study, subjects will come to TNO every week. Each of the four study periods will be performed identically.

In the first study period, on days -01, 07, 14, 21 and 28, subjects will come to TNO for collection of study substances for the coming week. On days 14, 21 and 28 they will come in a fasting state in the morning for blood sampling (fasting). Fasting blood samples will be taken by venapuncture.

After having received new study substances and the diary for the coming week, subjects can leave TNO.

On day 34, subjects will come to TNO at around 8:00 am and they will stay at TNO till about 11:00 for an oral glucose tolerance test. Fasting blood samples will be collected for determining treatment parameters. Subsequently subjects are provided the oral glucose load of 75 g glucose dissolved in 300 ml water. Blood samples will be taken at t= 90 and 120 min after the glucose load. After the last sample of the OGTT has been collected, subjects will be asked to void their bladder and afterwards receive a bottle for collection of 24 hour urine. The subjects will receive a free breakfast and can leave TNO.

The next day, on Day 35, subjects consume the breakfast as provided by TNO at home at around 8:00.They will come to TNO at around 11:00 am and they will stay at TNO till about 20:00. In addition, they will turn in the urine bottle after having voided their bladder at 24 after start of collection.

A canula will be inserted for collection of samples the rest of the day. At four hours after consumption subjects are provided a high fat meal. Blood samples will be taken at t = 30, 60, 120, 180, 240 and 360 min after the meal. Throughout the challenge sampling subjects are only allowed to drink water. After the last sample of the test has been taken subjects will receive a free dinner. After dinner an adipose tissue biopsy will be taken under local anesthesia.

The subjects will receive new study substances and diary for the coming week, starting on the next day.

In the next three study periods, the procedure will be identical.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the Health and lifestyle questionnaire Physical examination. Results of the pre-study laboratory tests
2. Males aged over 18 and < 60 years at Day 01 of the study
3. Body Mass Index (BMI): 26 - 35 (including) kg/m2
4. C-reactive protein (CRP) 1-10 mg/L. Acute inflammation as reason for increased CRP to be excluded based on white blood cell counts
5. Willing to use the study substances (yogurt and capsules) daily for 20 weeks
6. Normal Dutch eating habits as assessed by questionnaire
7. Voluntary participation and having given written informed consent
8. Willing to comply with the study procedures, including no use of food supplements, probiotic containing products and NSAID
9. Willing not to serve as blood donor during the study
10. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data
11. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
3. Having a chronic disease related to inflammation (such as arthritis) or a history of medical or surgical events that may significantly affect the study outcome, including diabetes (type 1 or 2) cardiovascular disease and hypothyroidemy
4. High blood pressure (age <55 y: DBP > 100 or SBP >160 mm Hg, age 55-59: DBP > 90 or SBP >140 mm Hg)
5. Fasting blood glucose level >6.9 mmol/L
6. Fasting cholesterol > 8 mmol/L
7. Blood hemoglobin < 8 mmol/L
8. Use of medication that might interfere with parameters to be measured or with one of the treatments
9. Frequent use of antibiotic medication (3 times or more in the past year)*
10. Frequent use of NSAID or paracetamol (frequency and/or urgency of need incompatible with participation - to be decided by medical investigator)
11. Lactose intolerance
12. Smoking
13. Extreme physical exercise > 6 hours/week
14. Reported unexplained weight loss or gain of > 4 kg in the month prior to the pre-study screening
15. Alcohol consumption > 28 units per week
16. Reported slimming or medically prescribed diet
17. Recent blood donation (< 1 month prior to the start of the study)
18. Personnel of TNO Quality of Life, their partner and their relatives in the first and second remove
19. Not having a general practitioner
20. Not willing to accept information transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
inflammation parameters | 5 weeks

SECONDARY OUTCOMES:
glucose and fat response | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gertruud Bakker, PhD, Principal Investigator — TNO Quality of Life, Zeist, The Netherlands
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands

REFERENCES:
- [Derived] Bakker GC, van Erk MJ, Pellis L, Wopereis S, Rubingh CM, Cnubben NH, Kooistra T, van Ommen B, Hendriks HF. An antiinflammatory dietary mix modulates inflammation and oxidative and metabolic stress in overweight men: a nutrigenomics approach. Am J Clin Nutr. 2010 Apr;91(4):1044-59. doi: 10.3945/ajcn.2009.28822. Epub 2010 Feb 24. PMID 20181810